CLINICAL TRIAL: NCT06995690
Title: Impact of Sub-anesthetic Dose of Ketamine in the Prevention of Post Spinal Hypotension in Patients Undergoing Orthopedic Surgeries
Brief Title: Ketamine for Preventing Post-Spinal Hypotension in Orthopedic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU MS 70/2025
Record Dates: First submitted 2025-05-21; First posted 2025-05-29 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Post-spinal Hypotension; Orthopedic Surgery; Spinal Aneshtesia
Keywords: Ketamine; Sub-anesthetic dose; Hypotension prevention; Neuraxial anesthesia; Hemodynamic stability; regional anesthesia; ASA I-II; Double-blind randomized trial; Blood pressure monitoring; Ephedrine use
MeSH Terms: interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine Group (Experimental): Patients receive crystalloid preloading of 15ml/kg (Ringer's lactate) +the sub-anesthetic dose of ketamine of 0.5 mg/kg IV added to the first bottle of ringer for blinding over 20 min before the spinal injection.
  Interventions: Drug: Ketamine
- Control Group (Placebo Comparator): Patients receive a crystalloid preloading of 15 ml/kg (Ringer's lactate)+ 0.5 mg/kg IV of Normal Saline added to the first bottle of ringer for blinding, over 20 min before the spinal injection.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ketamine — Patients receive crystalloid preloading of 15ml/kg (Ringer's lactate) +the sub-anesthetic dose of ketamine of 0.5 mg/kg IV added to the first bottle of ringer for blinding over 20 min before the spinal injection.
  Arms: Ketamine Group
Drug: Normal Saline — Patients receive a crystalloid preloading of 15 ml/kg (Ringer's lactate)+ 0.5 mg/kg IV of Normal Saline added to the first bottle of ringer for blinding, over 20 min before the spinal injection.
  Arms: Control Group

SUMMARY:
This randomized, double-blind, controlled clinical trial investigates the efficacy of a sub-anesthetic dose of ketamine (0.5 mg/kg IV) in preventing post-spinal hypotension in patients undergoing elective orthopedic surgeries under spinal anesthesia. The study compares ketamine with placebo (normal saline) in terms of blood pressure stability and incidence of hypotensive episodes following spinal anesthesia.

DETAILED DESCRIPTION:
Spinal anesthesia is commonly used for orthopedic procedures due to its effectiveness and favorable recovery profile. However, spinal-induced hypotension is a frequent complication resulting from sympathetic blockade, which can compromise organ perfusion and increase perioperative risk. This study aims to determine whether a single sub-anesthetic dose of intravenous ketamine administered before spinal anesthesia can reduce the incidence of hypotension.

Patients will be randomly allocated to either a ketamine group (receiving 0.5 mg/kg ketamine IV diluted in Ringer's lactate) or a control group (receiving volume-equivalent normal saline). Both interventions are administered over 20 minutes prior to the spinal injection to ensure blinding. All patients will undergo standard spinal anesthesia with 0.5% heavy bupivacaine plus fentanyl.

Primary outcome is the incidence of hypotension (defined as a mean arterial pressure drop >20% from baseline). Secondary outcomes include bradycardia, nausea, vomiting, hallucinations, and total dose of vasopressors required. The findings aim to support or refute the use of ketamine as a prophylactic strategy to stabilize hemodynamics during spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients American Society of Anesthesiologists Physical Status (ASA) I to II undergoing orthopedic surgeries under spinal anesthesia.
* Both Sexes.
* Patients aged equal to or above 18 years.
* Body mass index <35 kg/m2
* Duration of operation from 1 hour to 3 hours

Exclusion Criteria:

* Patients' refusal of procedure or participation in the study.
* Patients with contraindication to spinal anesthesia.
* Patients with cardiovascular or pulmonary disease.
* Patients with pre-procedural hypotension (systolic arterial pressure less than 90 mmHg and/or mean arterial pressure less than 60 mmHg).
* Patients aged below 18 years.
* Duration of operation below 1 hour or above 3 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Post-Spinal Hypotension | From spinal injection to end of surgery
  Hypotension is defined as a mean arterial pressure (MAP) less than 20% below baseline. MAP will be calculated using the formula: MAP = DBP + (SBP - DBP)/3.
  Hypotension will be treated with boluses of IV Ephedrine (3mg) and repeated if needed. The total dose of ephedrine required to correct hypotension and raise the MAP to the baseline will be recorded.

SECONDARY OUTCOMES:
Incidence of Hallucinations | From spinal injection to end of surgery
  Visual or auditory disturbances post ketamine administration. Midazolam (2 mg IV) will be given pre-injection to mitigate risk.
Incidence of Bradycardia | From spinal injection to end of surgery
  Bradycardia is defined as Heart Rate less than 50 beats per minute. Bradycardia will be treated with IV atropine (0.04 mg/kg) and repeated if needed.
Incidence of Nausea and Vomiting | From spinal injection to end of surgery
  Nausea is defined as an unpleasant subjective urge to vomit and Vomiting is defined as propulsive abdominal muscular spasms associated with the expulsion of gastric contents.
  Nausea and vomiting will be treated with 3 mg IV Granisetron.

CONTACTS AND LOCATIONS:
Overall Officials: Reem H El Kabarity, M.D, Principal Investigator — Faculty of Medicine, Ain Shams University
Locations (1):
- Ain Shams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
This is an academic study with a limited sample size, and there is no current plan to share de-identified participant data publicly.